CLINICAL TRIAL: NCT07133503
Title: Evaluation of Buccal Bone Thickness, Ridge Dimensions, And Root Position In Anterior Maxilla For Immediate Implant Placement
Brief Title: Radiological Evaluation of Anterior Maxilla For Immediate Implant Placement
Status: Completed | Type: Observational
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Duygu Kilic, Assistant professor, TC Erciyes University
Other Study IDs: EU2020/470
Record Dates: First submitted 2025-07-22; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Maxillary Retrusion
Keywords: Immediate implant applications; Cone-beam computed tomography; Anterior maxilla; Alveolar ridge morphology; Aging
MeSH Terms: conditions — Retrognathia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- 20-29 age group: In this age group bilateral central incisors, lateral incisors, and canines in the upper anterior region were examined
  Interventions: Other: radiological evaluation
- 30-39 age group: In this age group bilateral central incisors, lateral incisors, and canines in the upper anterior region were examined
  Interventions: Other: radiological evaluation
- 40-49 age group: In this age group bilateral central incisors, lateral incisors, and canines in the upper anterior region were examined
  Interventions: Other: radiological evaluation
- 50-59 age group: In this age group bilateral central incisors, lateral incisors, and canines in the upper anterior region were examined
  Interventions: Other: radiological evaluation
- 60-69 age group: In this age group bilateral central incisors, lateral incisors, and canines in the upper anterior region were examined
  Interventions: Other: radiological evaluation
- 70-80 age group: In this age group bilateral central incisors, lateral incisors, and canines in the upper anterior region were examined
  Interventions: Other: radiological evaluation

INTERVENTIONS:
Other: radiological evaluation — Using a line drawn through the midpoints of the teeth, parallel to their long axes, the anterior crest morphology was assessed. For maxillary central, lateral, and canine teeth, alveolar crest width and height, buccal bone thickness, and tooth-crest angle were measured separately. To determine buccal bone thickness, measurements were taken from the buccal crest apex, the midpoint of the root, and the apex of the tooth. The height of the alveolar crest was defined as the length of a line drawn parallel to the crest's long axis between the nasal fossa floor and the alveolar crest. The width of the alveolar crest was calculated by averaging measurements taken from the midpoints of three equal sections of the alveolar crest. The buccal undercut was determined as the point where the crest came closest to the root in the sagittal plane. Additionally, the angle between the tooth roots and the alveolar crest was measured to determine the root position in the radial plane

SUMMARY:
According to the literature age and gender may be associated with differences in skeletal size, anatomy and architecture in humans. However, little is known about the synergistic effects of age and gender on the healing capacity of maxillary bones, since most of the preclinical studies are focused on each variable separately. The present study radiologically evaluated various parameters such as alveolar crest height and width, buccal bone thickness, degree of buccal undercut, and root-crest angle using cone-beam computed tomography (CBCT) in a large patient population, and compared these parameters across different age and gender groups to analyze the effect of aging and gender on the bone morphology in the anterior maxillary region.

DETAILED DESCRIPTION:
Aim: The aim of this present study was to radiologically evaluate the socket morphology that may have a clinical impact on the outcomes of immediate implant placement in the anterior maxilla, using cone-beam computed tomography (CBCT) in a large patient population. Moreover, the parameters were compared between different age and gender groups to analyze the effect of aging and gender on the bone morphology around the maxillary anterior teeth.

Material and Methods: This study evaluated a total of 1,668 teeth in the esthetic region, including bilateral central incisors, lateral incisors, and canines in the upper anterior region, using CBCT images from 278 individuals. CBCT images were grouped into age ranges of 20-29, 30-39, 40-49, 50-59, 60-69, and 70-80 years. The morphology of the anterior ridge was assessed by separately measuring alveolar ridge width and height, buccal bone thickness, tooth-crest angle, and buccal undercut for maxillary central incisors.

ELIGIBILITY:
Inclusion Criteria:

-Between January 2015 and January 2024, undergoing CBCT imaging at the Erciyes University Faculty of Dentistry, Department of Oral and Maxillofacial Radiology

Exclusion Criteria:

* Systemic diseases,
* Anterior maxillary tooth loss,
* Having root canal treatments,
* Periapical lesions,
* History of or ongoing periodontal disease,
* Smoking.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cone-beam coemputed tomography (CBCT) images of individuals, obtained for various diagnostic purposes at the Erciyes University Faculty of Dentistry, Oral and Maxillofacial Radiology Clinic between January 2015 and January 2024
Sampling Method: Non-Probability Sample
Enrollment: 278 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Alveolar Crest Height | One year
  The height of the alveolar crest was defined as the length of a line drawn parallel to the crest's long axis between the nasal fossa floor and the alveolar crest.
Alveolar Crest Width | One year
  The width of the alveolar crest was calculated by averaging measurements taken from the midpoints of three equal sections of the alveolar crest.
Buccal Bone Thickness | One year
  To determine buccal bone thickness, measurements were taken from the buccal crest apex, the midpoint of the root, and the apex of the tooth.
Buccal Undercut Depth | One year
  The buccal undercut was determined as the point where the crest came closest to the root in the sagittal plane.
Root Position | One year
  the angle between the tooth roots and the alveolar crest was measured to determine the root position in the radial plane

CONTACTS AND LOCATIONS:
Overall Officials: Duygu Kilic, Study Director — TC Erciyes University
Locations (2):
- Turkey (Türkiye) (2):
  - Erciyes University Faculty of Dentistry Department of Periodontology, Kayseri, Kayseri̇
  - Erciyes University, Kayseri, Melikgazi

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-05-01): https://cdn.clinicaltrials.gov/large-docs/03/NCT07133503/Prot_SAP_000.pdf